CLINICAL TRIAL: NCT03775915
Title: The Use of Real-Time fMRI and a Mobile EEG System to Provide Neurofeedback to Stroke Patients to Promote Neural Plasticity for Motor Rehabilitation.
Brief Title: Neurofeedback for Stroke Rehabilitation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 lockdown and halt of clinical trials
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: StrokeNF
Record Dates: First submitted 2018-12-06; First posted 2018-12-14 (Actual); Results first posted 2021-08-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2020-07

CONDITIONS: Stroke
Keywords: Motor function; Brain activity
MeSH Terms: conditions — Stroke | interventions — Neurofeedback

STUDY DESIGN:
Intervention Model Description: Participants are randomly allocated (1:1 ratio) to either the intervention group (Real Neurofeedback) or the control group (Sham Neurofeedback). Randomisation is done after participants undergo baseline measurements using a computer-generated minimisation method that takes into account baseline upper limb function (Action Research Arm test score) and time since stroke.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real Neurofeedback (Experimental): 3 sessions of Real Neurofeedback over 1 week
  Interventions: Other: Neurofeedback
- Sham Neurofeedback (Sham Comparator): 3 sessions of Sham Neurofeedback over 1 week
  Interventions: Other: Sham Neurofeedback

INTERVENTIONS:
Other: Neurofeedback — A visual representation of the participants brain activity during movement of their affected hand in the MRI scanner.
  Arms: Real Neurofeedback
Other: Sham Neurofeedback — A visual representation of brain activity pre-recorded from a previous participant
  Arms: Sham Neurofeedback

SUMMARY:
Real-time neurofeedback aims to alter brain activation patterns through online feedback of ongoing brain activity using magnetic resonance imagining (MRI). Stroke survivors will be randomised to receive 3 sessions of real or sham neurofeedback. This study aims to investigate whether: 1) stroke survivors can maintain alterations in brain activity after the feedback is removed, 2) neurofeedback training leads to improvements in movement of the hand and arm, 3) neurofeedback training leads to changes in brain structure and function, 4) variability in response across people can be understood.

DETAILED DESCRIPTION:
Many stroke survivors experience impairment in upper limb function, reducing independence in activities of daily living. These impairments are associated with atypical brain activity patterns. Real-time neurofeedback aims to alter brain activation patterns through online feedback of ongoing brain activity using magnetic resonance imagining (MRI). Patterns of brain activity are displayed to a participant while a task is being performed. The participant is instructed to try to alter the patterns in a particular way, promoting specific brain activity patterns. Previous studies have found that people with and without stroke are capable of utilising the feedback to alter their brain activity. This study aims to investigate whether:

1. stroke survivors can maintain alterations in brain activity after the feedback is removed
2. neurofeedback training leads to improvements in movement of the hand and arm
3. neurofeedback training leads to changes in brain structure and function
4. variability in response across people can be understood.

30 stroke survivors (> 6 months after stroke), with residual upper limb impairment, will be recruited between February 2018 and December 2020. Participants will be randomised to receive 3 sessions of real or sham neurofeedback over one week, taking place at the Wellcome Centre for Integrative Neuroimaging, University of Oxford. Changes in brain activity during affected hand movements will be assessed with and without feedback using functional MRI and after feedback sessions using electroencephalography (EEG). Brain connectivity and structure will also be assessed using MRI at baseline and at a follow-up one week later. Clinical measures of upper limb function and impairment will be performed at baseline and at follow up sessions one week and one month later (Action Research Arm Test, Fugl-Meyer upper limb assessment, Jebsen Taylor hand function test), and in each session following neurofeedback (Jebsen taylor test).

ELIGIBILITY:
Inclusion Criteria:

* Stroke > 6 months previously
* Unilateral upper limb impairment, but physically able to complete the tasks required

Exclusion Criteria:

* Contraindications to MRI, such as a pacemaker, metallic implants or aneurysm clips
* Inability to provide informed consent
* Inability to actively participate in the research procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Johansen-Berg, PhD, Principal Investigator — University of Oxford
Locations (1):
- Wellcome Centre for Integrative Neuroimaging (WIN), Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymous data may be shared with other researchers on request
Supporting Information: Analytic Code
Time Frame: Analysis code may be shared following publication of the study results. There is no set end date for this
Access Criteria: Upon reasonable request to the PI

REFERENCES:
- [Derived] Sanders ZB, Fleming MK, Smejka T, Marzolla MC, Zich C, Rieger SW, Luhrs M, Goebel R, Sampaio-Baptista C, Johansen-Berg H. Self-modulation of motor cortex activity after stroke: a randomized controlled trial. Brain. 2022 Oct 21;145(10):3391-3404. doi: 10.1093/brain/awac239. PMID 35960166

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the community, between February 2018 and March 2020
Pre-assignment Details: 3 participants were not randomised to a group. 1 was withdrawn because the location of their stroke lesion made it impossible to deliver the intervention. 1 withdrew because they did not like the MRI scan. 1 was unable to continue due to study suspension because of the coronavirus pandemic.
Period: Overall Study
Arm/Group | Real Neurofeedback | Sham Neurofeedback
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Real Neurofeedback | Sham Neurofeedback | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (11) | 59 (13) | 62 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 8 | 11 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 12 | 12 | 24
Affected Hand [Count of Participants; unit: Participants] — Right, Left
  Participants
    Right | 2 | 6 | 8
    Left | 10 | 6 | 16
Time since stroke [Mean (Standard Deviation); unit: months] | 79 (70) | 72 (63) | 76 (65)

OUTCOME MEASURES:

1. Primary Outcome: Lateralisation of Brain Activity
Description: Lateralisation of brain activity during movement of the affected hand, assessed using functional magnetic resonance imaging (fMRI) blood oxygen level dependent (BOLD) signal. The activation in the region of interest is calculated for each hemisphere and the laterality index calculated as: (ipsilesional hemisphere - contralesional hemisphere) / (ipsilesional hemisphere + contralesional hemisphere). As such, positive values are indicative of greater activation in the ipsilesional hemisphere.
Time Frame: Throughout the 3 intervention sessions, an average of 4 days
Measure: Mean (95% Confidence Interval); unit: laterality index adjusted for baseline
Arm/Group | Real Neurofeedback | Sham Neurofeedback
Number analyzed (Participants) | 12 | 12
laterality index adjusted for baseline
  Day 2 | 0.23 [0.15 to 0.31] | 0.30 [0.22 to 0.39]
  Day 3 | 0.26 [0.17 to 0.34] | 0.22 [0.13 to 0.31]
  Day 4 | 0.25 [0.17 to 0.34] | 0.25 [0.16 to 0.34]
Statistical Analysis 1: Comparison: Real Neurofeedback vs Sham Neurofeedback; Test type: Other; p > 0.05, Linear Mixed Model — p-value calculated for interaction between group and day; Linear mixed effects model adjusted for baseline, F(2,46) = 1.061, p >0.05

2. Primary Outcome: Hand Function Assessed With the Jebsen Taylor Hand Function Test (Time, in Seconds)
Description: Performance on the Jebsen Taylor hand function test (time, in seconds to complete specified activities reflecting daily living)
Time Frame: Throughout study completion, 5 assessment sessions spread over approximately 3 weeks
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Real Neurofeedback | Sham Neurofeedback
Number analyzed (Participants) | 12 | 12
seconds
  Day1 | 267 (73) | 274 (77)
  Day2 | 238 (64) | 270 (77)
  Day3 | 221 (59) | 267 (75)
  Day4 | 220 (61) | 233 (64)
  Day5 | 214 (61) | 249 (70)
Statistical Analysis 1: Comparison: Real Neurofeedback vs Sham Neurofeedback; Test type: Superiority; p > 0.05, Mixed Models Analysis

3. Secondary Outcome: Change in Lateralisation of Brain Activity
Description: Change in lateralisation of brain activity during movement of the affected hand, assessed using functional magnetic resonance imaging (fMRI) blood oxygen level dependent (BOLD) signal.
Time Frame: 1 week follow up
Reporting Status: Not Posted

4. Secondary Outcome: Lateralisation of Brain Activity During Visuomotor Squeeze Task (MRI)
Description: Lateralisation of brain activity during a visuomotor squeeze task, assessed using functional magnetic resonance imaging (BOLD signal). The activation in the region of interest is calculated for each hemisphere and the laterality index calculated as: (ipsilesional hemisphere - contralesional hemisphere) / (ipsilesional hemisphere + contralesional hemisphere). As such, positive values are indicative of greater activation in the ipsilesional hemisphere.
Time Frame: Baseline, 1 week follow up
Population: Outliers removed on the basis of head motion or laterality index greater than 2 standard deviations from the mean
Measure: Mean (Standard Error); unit: laterality index
Arm/Group | Real Neurofeedback | Sham Neurofeedback
Number analyzed (Participants) | 10 | 9
laterality index
  Baseline | 0.31 (0.03) | 0.21 (0.06)
  1 week follow up | 0.29 (0.03) | 0.28 (0.05)

5. Secondary Outcome: Lateralisation of Brain Activity During Visuomotor Squeeze Task (EEG)
Description: Change in lateralisation of brain activity during a visuomotor squeeze task, assessed using EEG
Time Frame: Throughout study completion, an average of 3 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Upper Limb Function
Description: Action research arm test score (ARAT; upper limb function). Range 0-57, higher numbers indicate better upper limb function
Time Frame: Baseline, 1 week follow up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Real Neurofeedback | Sham Neurofeedback
Number analyzed (Participants) | 12 | 12
score on a scale
  Baseline | 31.9 (3.5) | 35.3 (3.9)
  1 week follow up | 34.3 (3.7) | 35.8 (3.7)

7. Secondary Outcome: Change in Upper Limb Function
Description: Change in action research arm test score (ARAT; upper limb function). Range 0-57, higher numbers indicate better upper limb function
Time Frame: 1 month follow up
Population: Only participants who were able to attend the 1 month follow up are included
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Real Neurofeedback | Sham Neurofeedback
Number analyzed (Participants) | 7 | 10
score on a scale
  Baseline | 31.7 (5.5) | 38.3 (3.9)
  1 month follow up | 34.7 (5.7) | 38.5 (3.4)

8. Secondary Outcome: Upper Limb Impairment
Description: Upper limb Fugl Meyer assessment score (upper limb impairment). Range 0-66, higher numbers indicate less upper limb impairment
Time Frame: Baseline, 1 week follow up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Real Neurofeedback | Sham Neurofeedback
Number analyzed (Participants) | 12 | 12
score on a scale
  Baseline | 44.2 (2.9) | 44.3 (4.0)
  1 week follow up | 45.8 (2.2) | 46.3 (3.5)

9. Secondary Outcome: Upper Limb Impairment
Description: as for outcome 8
Time Frame: Baseline, 1 month follow up
Population: Only participants who were able to attend the 1 month follow up are included
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Real Neurofeedback | Sham Neurofeedback
Number analyzed (Participants) | 7 | 10
score on a scale
  Baseline | 45.7 (3.9) | 46.2 (4.5)
  1 month follow up | 46.6 (3.9) | 47.7 (3.8)

10. Secondary Outcome: Change in Resting State Functional Connectivity
Description: Change in resting state functional connectivity, assessed using fMRI Analysis still in progress
Time Frame: 1 week follow up
Reporting Status: Not Posted, anticipated posting 2024-07

11. Secondary Outcome: Change in White Matter Tract Integrity
Description: Change in integrity of the white matter tracts, assessed using diffusion tensor imaging Analysis nearly completed
Time Frame: 1 week follow up
Reporting Status: Not Posted, anticipated posting 2024-07

12. Secondary Outcome: Change in Grey Matter Volume
Description: Change in grey matter volume derived from structural (T1) MRI Analysis still in progress
Time Frame: Baseline, 1 week follow up
Reporting Status: Not Posted, anticipated posting 2024-07

13. Secondary Outcome: Change in White Matter Microstructure
Description: Change in white matter microstructure, specifically myelin content, assessed using MRI Multi-Parameter Mapping
Time Frame: 1 week follow up
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Baseline Structure and Function as a Correlate of Response to Neurofeedback
Description: The correlation between baseline measures and change in lateralisation of brain activity during movement of the affected hand will be tested in order to identify markers to explain variability in response to real neurofeedback.
  Analysis still in progress
Time Frame: Throughout study completion, an average of 3 weeks.
Reporting Status: Not Posted, anticipated posting 2024-07

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Real Neurofeedback | Sham Neurofeedback
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
Early termination due to COVID leading to smaller numbers enrolled in the study than originally planned. Interim analysis at the stopping point revealed results that were deemed unlikely to change with additional participants and so the study was closed and full analysis is in progress.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT03775915/Prot_SAP_000.pdf